CLINICAL TRIAL: NCT01984307
Title: A Retrospective Swedish Cohort Study on Health Outcomes, Life Expectancy, Resource Use and Costs in Patients With a History of Myocardial Infarction and Additional Risk Factors for Atherothrombosis
Acronym: HELICON
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: ME-CV-1302
Record Dates: First submitted 2013-10-22; First posted 2013-11-14 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-05

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute coronary syndrome; Myocardial infarction; retrospective; cohort study; Healthcare resources utilization
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To characterize and estimate the size of different populations with a history of acute coronary syndrome in Sweden. To assess the burden of illness (co-morbidities, mortality rates healthcare resource utilization and atherothrombotic events) among patients with a history of myocardial infarction (MI) 1-3 years ago and additional risk factors for atherothrombosis.

ELIGIBILITY:
Inclusion Criteria:

- Patients hospitalised for ACS between 01.07.2006 and 31.06.2011.

Exclusion Criteria:

- Not applicable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with acute coronary syndrome with a history of MI 1-3 years ago.
Sampling Method: Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2013-08; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Description of study population in terms of death, cardiovascular disease events and health care resource utilization | Follow up period 1-7 years
  1. Death (all cause and CVD death) 2. CVD event (MI or Stroke) 3. Health care resource use and costs.
Assessment of the burden of illness among high risk patients with a history of MI | Follow up period 1-7 years
  1. Describe patients' demographics and clinical characteristics 2. Assess rate of CV event (MI and stroke), CV mortality and all cause mortality 3. Assess rate of CV events (MI and stroke), CV mortality and all cause mortality in patients having at least 24 months and 36 months without MI, respectively 4. Assess the impact of additional atherothrombotic risk factors 5. Describe treatment patterns 6. Evaluate healthcare resource use and costs 7. Assess predictors of new CV events (MI and stroke), CV mortality and all cause mortality
Assessment of the mortality rates among high risk patients with a history of MI | Follow up period 1-7 years
  1. Describe patients' demographics and clinical characteristics 2. Assess rate of CV event (MI and stroke), CV mortality and all cause mortality 3. Assess rate of CV events (MI and stroke), CV mortality and all cause mortality in patients having at least 24 months and 36 months without MI, respectively 4. Assess the impact of additional atherothrombotic risk factors 5. Describe treatment patterns 6. Evaluate healthcare resource use and costs 7. Assess predictors of new CV events (MI and stroke), CV mortality and all cause mortality

SECONDARY OUTCOMES:
Description of the high risk patient population in terms of CVD events, bleedings and co-morbidities. | Follow up period 1-7 years
  1. Assess rate of other CVD events (including heart failure, atrial fibrillation, angina pectoris) 2. Assess prevalence and rate of (major) organ specific bleedings (recorded diagnose in hospital) 3. Describe patients/proportions of patients with increased bleeding risk (history of previous bleedings, age, anti-thrombotic treatment etc) 4. Assess the prevalence of major co-morbidities in this population: (e.g. bradycardia, insertion of pacemaker, acute liver and renal failure) 5. To describe the death rate for the most common cause of deaths in the study population relative to the standardized death rate in the Swedish population and calculate the standardised mortality ratio

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Janzon, MD, PhD, Principal Investigator — Department of Cardiology, Linköping University Hospital, S-581 85 Linköping, Sweden
Locations (1):
- Research Site, Linköping, Sweden

REFERENCES:
- [Derived] Janzon M, Henriksson M, Hasvold P, Hjelm H, Thuresson M, Jernberg T. Long-term resource use patterns and healthcare costs after myocardial infarction in a clinical practice setting: results from a contemporary nationwide registry study. Eur Heart J Qual Care Clin Outcomes. 2016 Oct 1;2(4):291-298. doi: 10.1093/ehjqcco/qcw019. PMID 29474723